CLINICAL TRIAL: NCT00568893
Title: An Open Label Study of Drotrecogin Alfa (Activated) in Adult Patients With Severe Sepsis and Multiple Organ Dysfunctions A Phase IV Protocol
Brief Title: An Open Label Study of Severe Sepsis in Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7159; F1K-BX-S001
Record Dates: First submitted 2007-12-05; First posted 2007-12-06 (Estimated); Last update posted 2007-12-06 (Estimated); Status verified 2007-12

CONDITIONS: Severe Sepsis
MeSH Terms: conditions — Sepsis | interventions — drotrecogin alfa activated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): 24 microgram/kg/hr for 96 hours (+ or - 1 hour)
  Interventions: Drug: drotrecogin alfa (activated)

INTERVENTIONS:
Drug: drotrecogin alfa (activated)
  Other Names: LY203638; Xigris

SUMMARY:
This trial is to obtain safety data in adult patients with severe sepsis and two sepsis-induced organ infections who receive an infusion of drotrecogin alfa (activated).

DETAILED DESCRIPTION:
To collect safety data while providing drotrecogin alfa (activated) for the treatment of patients with severe sepsis with multiple organ dysfunctions. Patient access to drotrecogin alfa (activated) will be provided under this protocol prior to and during its review by the Authorities of Belgium and Luxemburg for commercial release.

ELIGIBILITY:
Inclusion Criteria:

* Patients greater than or equal 18 years of age may be included in this study only if they meet all of the following criteria:

  1. Must be 18 years.
  2. Suspected or proven infection
  3. Have or have had two or more sepsis-induced organ failures sepsis

Exclusion Criteria:

* Patients will be excluded from entry in this study for any of the following reasons:

  1. Documented first organ dysfunction greater than 48-hours prior to start of study drug.
  2. Patients greater than 135 kg in weight.
  3. Patients with a platelet count less than 30,000/mm3
  4. Active internal bleeding or at increased risk for bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2003-01; Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Safety Data | 9 Months

SECONDARY OUTCOMES:
All cause mortality data. | 9 Months
To determine the final disposition of sepsis patients treated with drotrecogin alfa (activated)(that is, patient location at discharge from study hospital or 90 days). | 9 Months

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (18):
- Belgium (18):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Antwerp
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arlon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bonheiden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bruges
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brussels
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ghent
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haine-St. Paul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hasselt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Huy
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Louvière
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leuven
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liège
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mons
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montigny-le-Tilleul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ottignies
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Roeselare
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Verviers
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wilrijk

REFERENCES:
- [Derived] Hodder RV, Hall R, Russell JA, Fisher HN, Lee B. Early drotrecogin alpha (activated) administration in severe sepsis is associated with lower mortality: a retrospective analysis of the Canadian ENHANCE cohort. Crit Care. 2009;13(3):R78. doi: 10.1186/cc7893. Epub 2009 May 20. PMID 19457240
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com